CLINICAL TRIAL: NCT00542425
Title: A Randomized, Parallel-Group, Phase 2 Dose-finding Study to Evaluate the Effects of BA058 in the Treatment of Postmenopausal Women With Osteoporosis
Brief Title: Phase 2 Dose-finding Study to Evaluate the Effects of BA058 in the Treatment of Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BA058-05-002
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Results first posted 2010-07-29 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-09

CONDITIONS: Osteoporosis
Keywords: osteoporosis; postmenopausal; bone loss
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Teriparatide; abaloparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BA058 20 µg (Experimental)
  Interventions: Drug: BA058 20 µg
- BA058 40 µg (Experimental)
  Interventions: Drug: BA058 40 µg
- BA058 80 µg (Experimental)
  Interventions: Drug: BA058 80 µg
- teriparatide (Active Comparator)
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: teriparatide — teriparatide 20 µg subcutaneous daily
  Other Names: PTH
  Arms: teriparatide
Drug: Placebo — Placebo subcutaneous daily
  Arms: Placebo
Drug: BA058 20 µg — BA058 20 µg subcutaneous daily
  Arms: BA058 20 µg
Drug: BA058 40 µg — BA058 40 µg subcutaneous daily
  Arms: BA058 40 µg
Drug: BA058 80 µg — BA058 80 µg subcutaneous daily
  Arms: BA058 80 µg

SUMMARY:
The purpose of this study is to determine whether BA058 is effective in building bone in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
This is a randomized, parallel-group, multi-center, dose-finding study to evaluate the effects of BA058 in the treatment of otherwise healthy postmenopausal women with osteoporosis.

ELIGIBILITY:
Primary Inclusion Criteria:

* The patient has a bone mineral density T-score ≤ 2.5 at the lumbar spine or hip (femoral neck) by dual energy x-ray absorptiometry (DXA). Women with a bone mineral density T-score of 2.0 or lower and a prior low-trauma forearm, humerus, vertebral, sacral, pelvic, hip, femoral, or tibial fracture within the past 5 years, or who have an additional risk factor such as age 65 or greater or a strong maternal history of osteoporosis defined as a fracture related to osteoporosis or osteoporosis itself as determined by BMD criteria, are also study candidates.
* The patient is in good general health as determined by medical history and physical examination and is without evidence of clinically significant abnormality in the opinion of the Investigator.

Primary Exclusion Criteria:

* History of bone disorders (e.g., Paget's disease) other than postmenopausal osteoporosis.
* Prior treatment with approved or as yet unapproved bone-acting investigational agents.
* History of carcinoma, nephrolithiasis or urolithiasis within the past five years or osteosarcoma at any time.
* History of radiotherapy (radiation therapy).

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Radius Health, Inc.
Locations (1):
- Radius Health, Inc., Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Leder BZ, O'Dea LS, Zanchetta JR, Kumar P, Banks K, McKay K, Lyttle CR, Hattersley G. Effects of abaloparatide, a human parathyroid hormone-related peptide analog, on bone mineral density in postmenopausal women with osteoporosis. J Clin Endocrinol Metab. 2015 Feb;100(2):697-706. doi: 10.1210/jc.2014-3718. Epub 2014 Nov 13. PMID 25393645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study started in the US, in January 2007. For the initial 24-week treatment period, patients were randomized to study treatment at 30 study centers in the US, Argentina, India and the UK . Eleven of the 30 study centers treated patients in the 24-week treatment extension period in the US, Argentina, and India.
Pre-assignment Details: After eligibility was established, patients entered a 4-week Pretreatment Period during which they received daily Calcium and Vitamin D supplements, were trained in self-injection with the pen devices, and were assessed for additional evaluations at the end of the Pretreatment Period. Patients who remained eligible were randomized on Day 1.
Period: Initial 24 Weeks
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide
Started | 46 | 43 | 43 | 45 | 45
Completed | 42 | 33 | 36 | 34 | 39
Not Completed | 4 | 10 | 7 | 11 | 6
Not completed — Administrative reasons | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 3 | 2
Not completed — Inability to complete procedures | 0 | 3 | 2 | 1 | 2
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Refusal of treatment | 2 | 2 | 1 | 4 | 1
Not completed — Other | 0 | 2 | 1 | 0 | 0
Period: Extended 24 Weeks of Treatment
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide
Started | 11 (Not all patients were eligible for extension study, often due to the regulatory approval timeline.) | 13 (Not all patients were eligible for extension study, often due to the regulatory approval timeline.) | 10 (Not all patients were eligible for extension study, often due to the regulatory approval timeline.) | 7 (Not all patients were eligible for extension study, often due to the regulatory approval timeline.) | 14 (Not all patients were eligible for extension study, often due to the regulatory approval timeline.)
Completed | 10 | 11 | 8 | 6 | 13
Not Completed | 1 | 2 | 2 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Refusal of treatment | 0 | 1 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide | Total
Number analyzed (Participants) | 46 | 43 | 43 | 45 | 45 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.11) | 66.3 (6.96) | 64.5 (7.35) | 64.8 (7.21) | 64.5 (7.48) | 65 (7.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 43 | 43 | 45 | 45 | 222
  Male | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Marker of Bone Metabolism, PINP
Description: PINP, N-terminal propeptide of type I procollagen, is a marker of anabolic bone growth.
Time Frame: 6 months
Population: The intent to treat (ITT) population included any patient who received at least one dose of study medication; N=221. 193 of the 221 ITT patients had data available for analysis at Week 24.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide
Number analyzed (Participants) | 38 | 34 | 37 | 42 | 42
Percent change from baseline | -13.1 (26.47) | 20.0 (61.05) | 90.8 (116.92) | 97.2 (123.88) | 154.3 (213.07)
Statistical Analysis 1: Comparison: Placebo vs BA058 40 µg; Study size provided 95 percent power to detect a difference in means of 114 (ng/mL) for PINP endpoint between BA058 (SD=147.5) and placebo (SD=34.5). Study size was based on Bauer 2006 data and utilized a 2-tailed 2-sample t-test with a significance level of alpha=0.01 with a Bonferonni adjustment for multiple testing. It included a 10 percent adjustment for within study dropouts over 6 months and a 15 percent adjustment to maintain adequate power for a per protocol analysis of key endpoints; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Placebo vs BA058 80 µg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

2. Primary Outcome: Change in Bone Mineral Density, Total Spine.
Description: Total analyzable spine bone mineral density (BMD) was analyzed by DXA at Week 24.
Time Frame: 6 months
Population: The intent to treat (ITT) population included any patient who received at least one dose of study medication; N=221. 187 of the 221 ITT patients had data available for analysis at Week 24.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide
Number analyzed (Participants) | 42 | 32 | 37 | 36 | 40
Percent change from baseline | 1.22 (3.211) | 3.30 (2.068) | 5.21 (4.427) | 6.11 (3.744) | 5.47 (4.218)
Statistical Analysis 1: Comparison: Placebo vs BA058 40 µg; For the BMD endpoint, the planned study size has 80 percent power with alpha=0.02 to detect a difference in mean change from baseline of 3.0 (percent) in BMD for the BA058 group and the BA058 Placebo group using an assumed SD of 3.5-4.0. The estimates for SD are based upon results of lumbar spine BMD presented by Body 2002; Test type: Superiority or Other; p < 0.001, ANOVA
Statistical Analysis 2: Comparison: Placebo vs BA058 80 µg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA

3. Secondary Outcome: Change in Bone Mineral Density, Femoral Neck.
Description: Femoral neck bone mineral density (BMD) was analyzed by DXA at Week 24.
Time Frame: 6 months
Population: The intent to treat (ITT) population included any patient who received at least one dose of study medication; N=221. 182 of the 221 ITT patients had data available for analysis at Week 24.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide
Number analyzed (Participants) | 41 | 31 | 37 | 35 | 38
Percent change from baseline | 0.79 (4.797) | 2.69 (4.022) | 2.20 (4.406) | 3.07 (4.175) | 1.07 (4.564)

4. Secondary Outcome: Change in Bone Mineral Density, Total Hip.
Description: Total analyzable hip bone mineral density (BMD) was analyzed by DXA at Week 24.
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide
Number analyzed (Participants) | 41 | 31 | 37 | 35 | 38
Percent change from baseline | 0.39 (3.053) | 1.43 (2.639) | 1.97 (3.699) | 2.60 (3.488) | 0.45 (3.925)

5. Secondary Outcome: Change in Bone Mineral Density, Total Spine.
Description: Total analyzable spine bone mineral density (BMD) was analyzed by DXA at Week 48.
Time Frame: 12 months
Population: The extension population included any patient who continued in the extended 24 weeks of treatment; N=55. 49 of the 55 extension patients had data available for analysis at Week 48.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide
Number analyzed (Participants) | 10 | 11 | 9 | 6 | 13
Percent change from baseline | 0.74 (3.541) | 5.14 (3.164) | 9.84 (5.313) | 12.94 (3.251) | 8.63 (6.8)

ADVERSE EVENTS:
Time Frame: For patients treated during the initial 6 months only, AEs were collected for 8 months (1 pre + 6 treatment + 1 post). For patients treated over the extended treatment period of 12 months, AEs were collected for 14 months (1 pre + 12 treatment + 1 post).
Description: Method of routinely determining whether or not certain adverse events have occurred was by regular investigator assessment and regular laboratory testing.
Arm/Group | Placebo | BA058 20 µg | BA058 40 µg | BA058 80 µg | Teriparatide
Serious Adverse Events (participants affected / at risk) | 1/45 | 2/43 | 0/43 | 2/45 | 0/45
Other Adverse Events (participants affected / at risk) | 30/45 | 31/43 | 32/43 | 33/45 | 35/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | BA058 20 µg (N=43) | BA058 40 µg (N=43) | BA058 80 µg (N=45) | Teriparatide (N=45)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bilateral crural hernia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=45) | BA058 20 µg (N=43) | BA058 40 µg (N=43) | BA058 80 µg (N=45) | Teriparatide (N=45)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 5 | 3 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 5 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 3 | 2 | 1 | 1
Injection site hematoma (General disorders) | 5 | 2 | 5 | 1 | 6
Injection site hemorrhage (General disorders) | 0 | 0 | 0 | 1 | 3
Bronchitis (Infections and infestations) | 1 | 3 | 2 | 3 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 3 | 0
Influenza (Infections and infestations) | 7 | 1 | 3 | 5 | 6
Nasopharyngitis (Infections and infestations) | 2 | 5 | 2 | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 4 | 1 | 1 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 2 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 5 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 6 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 6 | 6 | 6
Sciatica (Nervous system disorders) | 0 | 0 | 3 | 1 | 0
Hypercalciuria (Renal and urinary disorders) | 4 | 3 | 2 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI/Institution may publish/present results of the Study provided that the Publication is reviewed by the Sponsor for Confidential Information at least 60 days prior to submission. If the Publication contains patent-related information, the submission shall be delayed for 90 days.

The Institution/PI will not publish until after the data from the multi-center study is published in a combined paper as long as it is completed within 18 months from the date of study completion.